CLINICAL TRIAL: NCT03444480
Title: A Phase Ⅰb Study Evaluating the Pharmacokinetic,Safety and Efficacy of Remimazolam Tosylate in Healthy Volunteers
Brief Title: A Phase Ⅰb Study of Remimazolam Tosylate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RMZL-PIb
Record Dates: First submitted 2015-08-04; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — 4-methylbenzenesulfonic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remimazolam Tosylate 1 (Experimental): IV bolus of Remimazolam Tosylate with a loading dose of 0.4mg/kg body weight over 1 minute followed by a maintenance dose of 1.5mg/kg/h over 2 hours.1 h 55 min after dosing start， 0.5 mg Flumazenil is administered
  Interventions: Drug: Remimazolam Tosylate
- Remimazolam Tosylate 2 (Experimental): IV bolus of Remimazolam Tosylate with a loading dose of 0.4mg/kg body weight over 1 minute followed by a maintenance dose of 1.5mg/kg/h over 2 hours.1 h 55 min after dosing start time,0.5ml placebo is administered
  Interventions: Drug: Remimazolam Tosylate

INTERVENTIONS:
Drug: Remimazolam Tosylate — Initial dose plus supplemental doses
  Other Names: HR7056

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics/Pharmacodynamics and safety of Remimazolam Tosylate in healthy volunteers after loading/maintenance dose regimen.

DETAILED DESCRIPTION:
1. Study the Pharmacokinetics/Pharmacodynamics of Remimazolam Tosylate in healthy volunteers after loading/maintenance dose regimen.
2. Study the reversal effect and time required of Flumazepine on Rimazolam'effect.
3. Study the Safety of Remimazolam Tosylate in healthy volunteers after loading/maintenance dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤55 years.
* Weight range 50 to 100 kg and body mass index (BMI) 18 to 26 kg/m2.
* Willing and able to comply with the requirements of the protocol.
* Provide written informed consent to participate in the study.

Exclusion Criteria:

* Abnormal results of physical or laboratory examination with clinical significance
* With a history of laboratory results that show the presence of hepatitis B surface antigen (HBs Ag), hepatitis C antibody (HCV Ab), or human immunodeficiency virus (HIV).
* With evidence of uncontrolled renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic dysfunction, in the opinion of the investigator or medical monitor.
* Subject with clinically significant abnormalities in baseline 12-lead electrocardiogram (ECG) or vital signs（SBP <90 mmHg or >140 mmHg，DBP <50 mmHg or >90 mmHg；Hr <50 bpm or >100 bpm；SpO2 <95%）.
* Has a known sensitivity to benzodiazepines, flumazenil, or anesthetic agents, or a medical condition such that these agents are contraindicated.
* Receipt of other medication within 14 days of the first study day.
* Blood donation greater than 200 ml or participation in a clinical study of an unlicensed drug in the previous 3 months.
* History of smoking or alcohol abuse within 6 months of screening.
* History of grapefruit juice or any other foods affect the activity of cytochrome P450 3A4（CYP3A4） within 7 days of screening.
* Pregnant,lactating.
* Mallampati score ≥3.
* Patients who in the opinion of the investigator may not be able to comply with the requirements of the study are not eligible

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2014-08-16 (Actual); Study Completion 2014-08-16 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Remimazolam in human plasma. | From prior to study drug injection until 4 hours post-dose
Area under the plasma concentration versus time curve (AUC) of Remimazolam in human plasma. | From prior to study drug injection until 4 hours post-dose
Peak Plasma Concentration (Cmax) of M01 in human plasma. | From prior to study drug injection until 4 hours post-dose
  M01 is the main metabolite of Remimazolam
Area under the plasma concentration versus time curve (AUC) of M01 in human plasma. | From prior to study drug injection until 4 hours post-dose
  M01 is the main metabolite of Remimazolam

SECONDARY OUTCOMES:
Safety by measurement of Adverse Events. | From start of study drug injection to patient discharge (approx. 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Pei Hu, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen X, Sang N, Song K, Zhong W, Wang H, Jiang J, Huang Y, Hu P. Psychomotor Recovery Following Remimazolam-induced Sedation and the Effectiveness of Flumazenil as an Antidote. Clin Ther. 2020 Apr;42(4):614-624. doi: 10.1016/j.clinthera.2020.02.006. Epub 2020 Mar 13. PMID 32178858